CLINICAL TRIAL: NCT06444529
Title: A Double-Masked Comparison of Apraclonidine Hydrochloride Ophthalmic Solution to Vehicle for the Reduction of Ocular Redness
Brief Title: A Double-Masked Comparison of FID 123320 Ophthalmic Solution to Vehicle for the Reduction of Ocular Redness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DEW422-C001
Record Dates: First submitted 2024-05-31; First posted 2024-06-05 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Ocular Redness
Keywords: Eye redness; Irritated eyes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apraclonidine Hydrochloride Ophthalmic Solution (Experimental): One drop in each eye on Day 1, followed by 2 drops in each eye on Day 2 onward for approximately 8 weeks
  Interventions: Drug: Apraclonidine Hydrochloride Ophthalmic Solution
- Vehicle (Placebo Comparator): One drop in each eye on Day 1, followed by 2 drops in each eye on Day 2 onward for approximately 8 weeks
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Apraclonidine Hydrochloride Ophthalmic Solution — Investigational ophthalmic solution applied topically to the eye with a dropper bottle
  Other Names: FID 123320
  Arms: Apraclonidine Hydrochloride Ophthalmic Solution
Drug: Vehicle — Vehicle (inactive ingredients) applied topically to the eye with a dropper bottle
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Apraclonidine Hydrochloride Ophthalmic Solution 0.125% when compared to Vehicle, in relieving redness of the eye due to minor eye irritations. This study will be conducted in the United States.

DETAILED DESCRIPTION:
The study will consist of six (6) scheduled visits: Screening and/or Baseline Visit (Day -7 to -1), Eligibility Confirmation/Randomization/1st Treatment Visit (Day 1), Week 2 Follow-Up Visit (Day 14), Week 4 Follow-Up Visit (Day 28), Week 8 Follow-Up/Treatment Discontinuation Visit (Day 56) and Exit Visit (Day 63). The expected individual duration of participation in the study is approximately 10 weeks with approximately 56 days of exposure to the investigational product.

ELIGIBILITY:
Key Inclusion Criteria:

* Capable of giving signed informed consent;
* Willing and able to follow all instructions and attend all study visits;
* Able to self-administer eye drops- in the opinion of the investigator;
* History of redness relief drop use within the last 6 months, or a desire to use over-the-counter (OTC) eye drops for redness relief;
* Females capable of becoming pregnant: Agree to urine pregnancy tests and the use of medically acceptable forms of birth control throughout the study;
* Ocular health within normal limits, including best-corrected visual acuity (BCVA) of 20/40 or better in each eye as measured using a Snellen chart;
* Ocular redness at baseline as specified in the protocol;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Known contraindications or sensitivities to the use of any of the investigational drug(s) or their components, or any other medication required by the protocol;
* Ocular surgical interventions within 6 months prior to Visit 1 or during the study;
* Ocular conditions that, in the opinion of the investigator, could affect the subject's safety or study parameters (i.e., could affect ocular redness, intraocular pressure, or eyelid position);
* Disallowed medications or devices as specified in the protocol;
* Planned surgery (ocular or systemic) during the study period or within 30 days after the study period;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in investigator-assessed ocular redness at 15 minutes post-instillation on Day 1 | Day 1: Pretreatment; 15 minutes post-treatment
  Ocular redness will be assessed by the investigator using a scale from 0 to 4 in half-unit increments (0=none; 4=extremely severe). This endpoint is co-primary with the 10 hours post-instillation endpoint.
Mean change from baseline in investigator-assessed ocular redness at 10 hours (600 minutes) post-instillation on Day 1 | Day 1: Pretreatment; 10 hours (600 minutes) post-treatment
  Ocular redness will be assessed by the investigator using a scale from 0 to 4 in half-unit increments (0=none; 4=extremely severe). This endpoint is co-primary with the 15 minutes post-instillation endpoint.

SECONDARY OUTCOMES:
Mean change from baseline in investigator-assessed ocular redness at 1 minute post-instillation on Day 1 | Day 1: Pretreatment; 1 minute post-treatment
  Ocular redness will be assessed by the investigator using a scale from 0 to 4 in half-unit increments (0=none; 4=extremely severe).
Mean change from baseline in investigator-assessed ocular redness at 8 hours (480 minutes) post-instillation on Day 1 | Day 1: Pretreatment; 8 hours (480 minutes) post-treatment
  Ocular redness will be assessed by the investigator using a scale from 0 to 4 in half-unit increments (0=none; 4=extremely severe).
Mean change from baseline in investigator-assessed ocular redness at 12 hours (720 minutes) post-instillation on Day 1 | Day 1: Pretreatment; 12 hours (720 minutes) post-treatment
  Ocular redness will be assessed by the investigator using a scale from 0 to 4 in half-unit increments (0=none; 4=extremely severe).

CONTACTS AND LOCATIONS:
Overall Officials: Principal Clinical Trial Lead, Pharma, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Global Research Management, Glendale, California
  - Oculus Research, Inc., Garner, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Emerson Clinical Research Institute, Inc., Falls Church, Virginia
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No